CLINICAL TRIAL: NCT03905902
Title: A Phase III, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of DCVAC/OvCa Added to Standard of Care in Patients With Relapsed Platinum-sensitive Ovarian, Fallopian Tube, and Primary Peritoneal Carcinoma
Brief Title: DCVAC/OvCa and Standard of Care (SoC) in Relapsed Ovarian, Fallopian Tube, and Primary Peritoneal Carcinoma
Acronym: VITALIA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision
Sponsor: SOTIO a.s. (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOV09; VITALIA/ ENGOT-ov53 (Other: ENGOT)
Record Dates: First submitted 2019-04-02; First posted 2019-04-08 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Carcinoma
Keywords: active cellular immunotherapy; dendritic cells; platinum-sensitive; relapsed ovarian cancer; biologic
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Intervention Model Description: parallel-group, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCVAC/OvCa with standard of care (Experimental): Induction period: DCVAC/OvCa with carboplatin and gemcitabine, or carboplatin and paclitaxel, or carboplatin and pegylated liposomal doxorubicin, with or without bevacizumab
  Maintenance period: DCVAC/OvCa with bevacizumab, best supportive care or a PARPi
  Interventions: Biological: DCVAC/OvCa; Biological: DCVAC/OvCa placebo
- Placebo with standard of care (Placebo Comparator): Induction period: DCVAC Placebo with carboplatin and gemcitabine, or carboplatin and paclitaxel, or carboplatin and doxorubicin, with or without bevacizumab
  Maintenance Period:DCVAC placebo with bevacizumab, best supportive care or a PARPi carboplatin and gemcitabine or carboplatin and paclitaxel with or without bevacizumab, best supportive care or a PARPi
  Interventions: Biological: DCVAC/OvCa; Biological: DCVAC/OvCa placebo

INTERVENTIONS:
Biological: DCVAC/OvCa — activated autologous dendritic cells
  Other Names: dendritic cell vaccine/ ovarian cancer
Biological: DCVAC/OvCa placebo — placebo for activated autologous cells

SUMMARY:
Multi-center, phase III trial of DCVAC/OvCa added to standard of care treatments for relapsed ovarian cancer. Patients will receive study treatment until all doses are administered, or other criteria are met.

DETAILED DESCRIPTION:
All patients who meet entry criteria will be randomized, and will undergo a leukapheresis procedure. During the Induction period, all patients will receive DCVAC/OvCa or placebo (study treatment) with concurrent standard-of-care platinum-based chemotherapy, with or without use of bevacizumab. In the Maintenance period, patients will continue treatment with study treatment in combination with bevacizumab, a poly (ADP-ribose) polymerase inhibitor (PARPi) or best supportive care only. Study treatment will continue irrespective of disease progression

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade serous or endometrioid carcinoma of the ovary, peritoneum or fallopian tube.
* Without disease progression during preceding platinum-based chemotherapy
* Platinum-sensitive patients defined as Platinum-Free Interval of more than 6 months between the end of the last cycle of platinum-based chemotherapy and radiologic evidence of progression.
* First relapse identified by the criteria above up to 28 days prior to study randomization
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Known BRCA (breast cancer susceptibility gene) mutation status before randomization
* Patient is intended to be treated with bevacizumab, best supportive care (BSC) only or PARPi

Exclusion Criteria:

* Tumor-specific: any other histology sub-type that is not high grade serous or endometrioid, however a combination of these is allowed
* Disease Treatment history: started or ongoing systemic treatment for current relapse of Epithelial Ovarian Cancer, Fallopian Tube Cancer or Primary Peritoneal Cancer before signing informed consent form (ICF), concomitant use of anti-neoplastic anti- hormonal therapy
* Intention to treat with intra-peritoneal chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Overall Survival(OS) | Assessed from enrolment up to study completion, approximately 6.6 years
  Defined as the time from randomization until the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Assessed from enrollment to up to 4 years
  Defined as the time from randomization to the earlier date of objective progression or death due to any cause in the absence of progression.
Objective Response Rate | Assessed from start of treatment to up to 4 years
  Assessment of Objective Response Rate per RECIST1.1 until objective progression as defined by the Investigator.
Time to Relapse | Assessed from start of treatment up to 4 years
  Assessment of Time to Relapse, per objective progression according to RECIST 1.1.
Duration of Response | Assessed from start of study treatment up to 4 years
  Assessment of Duration of Response until objective progression per RECIST 1.1.
Biological Progression-Free Survival | Assessed from randomization up to study completion up to 6.6 years.
  Defined as the time from randomization to the earlier date of assessment of biological progression evaluated by increasing CA 125 levels or death due to any cause in the absence of progression.
Safety Assessments: NCI CTCAE version 5.0 | Assessed from Screening through 30 days after the completion of Investigational Medicinal Product approximately 18 months.
  Defined as the incidence, severity and outcome of treatment emergent adverse events (TEAEs), and serious adverse events (SAEs) assessed by NCI CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Fricke, MD PhD, Study Director — SOTIO a.s.; David Cibula, Prof. MD PhD, Principal Investigator — The Central and Eastern European Gynecologic Oncology Group

IPD SHARING:
Plan to Share IPD: Undecided